CLINICAL TRIAL: NCT00837915
Title: Comparative, Randomized, Single-Dose, Fully Replicated, 4-Way Crossover Bioavailability Study of Ranbaxy and Schering (Claritin_D® 24 Hour) Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets, in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Bioequivalnce Study of Loratadine / Pseudoephedrine Sulfate 10/ 240 mg Extended-Release Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA01111
Record Dates: First submitted 2009-01-08; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Bioequivaelnce Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended Release Tablets
MeSH Terms: interventions — Loratadine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets of Ranbaxy
  Interventions: Drug: Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets
- 2 (Active Comparator): (Claritin-D® 24 hour) Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets
  Interventions: Drug: Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets

INTERVENTIONS:
Drug: Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Ranbaxy and Schering (Claritin-D® 24 hour) Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets, in a fully replicated design, under fasting conditions.

DETAILED DESCRIPTION:
The study was conducted as an open-label, randomized, Single-Dose, Fully replicated, 4-way Crossover Study to compare the single-dose relative bioavailability of Ranbaxy and Schering (Claritin_D® 24 hour) Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets, in Healthy adult Volunteers Under Fasting Conditions A total of 40 subjects (30 males and 10 females) were included in this study, of which 36 (27 males and 9 females) finished the study according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers, 18-45 years of age
* Weighing at least 60 kg for males and 52 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983);
* Medically healthy subjects with clinically normal laboratory profiles;
* Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the study and throughout the study or be using one of the following acceptable birth control methods:

  * surgically sterile (bilateral tubal ligation, hysterectomy bilateral oophorectomy) 6 months minimum
  * IUD in place for at least 3 months
  * barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the start of the study and .throughout the study
  * surgical sterilization of the partner (vasectomy for 6 months minimum
  * hormonal contraceptives for at least 3 months prior to the start of the study
* Other birth control methods may be deemed acceptable.
* Postmenopausal women with amenorrhea for at least 2 years will be eligible;
* Voluntarily consent to participate in the study.

Exclusion Criteria:

* Subject candidates must not be enrolled in the study if they meet any of the following criteria:
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic,gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:

  * alcoholism or drug abuse within the past year
  * hypersensitivity or idiosyncratic reaction to loratidine or any other H1-receptor antagonist
  * hypersensitivity or idiosyncratic reaction to pseudoephederine or any other sympatomimetic amines
  * glaucoma or hypermetropia
* Subjects receiving a monoamine oxidase (MAO) inhibitor or within 14 days of stopping use of an MAO inhibitor, or any sympathomimetic amines.
* Subjects who have used any drugs or other substances known to be strong inhibitors of CYP (cytochrome P450) enzymes within 10 days of study start.
* Subjects who have used any drugs or other substances known to be strong inducers of CYP (cytochrome P450) enzymes within 28 days of study start.
* Female subjects who are pregnant or lactating.
* Subjects who have been on an abnormal diet (for whatever reason) during the 28 days prior to the first dose.
* Subjects who, through completition of the study, would have donated in excess of:

  * 500 mL of blood in 14 days, or
  * 500-750 mL of blood in 14 days (unless approved by the principal Investigator),
  * 1000 mL of blood in 90 days,
  * 1250 mL of blood in 120 days,
  * 1500 mL of blood in 180 days,
  * 2000 mL of blood in 270 days,
  * 2500 mL of blood in 1 days,
* Subjects who have participated in another clinical trial within 28 days prior to the study start.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-06; Primary Completion 2002-08 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability between Ranbaxy and Schering (Claritin-D® 24 hour) Loratadine 10mg /Pseudoephedrine Sulfate 240 mg Extended-Release Tablets under fasting conditions

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Montreal, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html